CLINICAL TRIAL: NCT01937793
Title: Swallowing Exercises for Patients With Nasopharyngeal Cancer After Radiation Therapy
Brief Title: Swallowing Exercises for Nasopharyngeal Cancer After Radiation Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201211062RIB; 000766KJY (Other: National Taiwan University Hospital)
Record Dates: First submitted 2013-01-30; First posted 2013-09-10 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Nasopharyngeal Cancer; Dysphagia
Keywords: radiation; speech-language pathology
MeSH Terms: conditions — Nasopharyngeal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- effortful swallowing exercise (Active Comparator): Subjects in the arm are asked to do the effortful swallowing exercise at home for 8 weeks. The training frequency is to exercise 3-4 days/week, 3 times/day, 10 repetitions per time. Besides the at home exercise, each subject is scheduled to meet the investigator at the hospital at weekly basis to discuss and review his/her exercise practice.
  Interventions: Other: effortful swallowing exercise
- Mendelsohn swallowing exercise (Active Comparator): Subjects in the arm are asked to do the Mendelsohn swallowing exercise at home for 8 weeks. The training frequency is to exercise 3-4 days/week, 3 times/day, 10 repetitions per time. Besides the at home exercise, each subject is scheduled to meet the investigator at the hospital at weekly basis to discuss and review his/her exercise practice.
  Interventions: Other: Mendelsohn swallowing exercise

INTERVENTIONS:
Other: effortful swallowing exercise — voluntarily increases the posterior tongue base pushing effort while swallowing
  Arms: effortful swallowing exercise
Other: Mendelsohn swallowing exercise — voluntarily increase the extent and duration of laryngeal elevation while swallowing
  Arms: Mendelsohn swallowing exercise

SUMMARY:
This study is designed to investigate the treatment efficacy of 8 weeks swallowing exercise programs for patients with NPC after radiation therapy. This study also compares two different swallowing exercise: effortful swallow and Mendelsohn's maneuver, to see which one can bring more benefits to patients after a certain period of exercise training. Three assessment tools are selected to evaluate the study result: Mann Assessment of Swallowing Ability (MASA), videofluoroscopic swallowing study (VFSS), and Chinese version Swallowing Quality-of-Life Questionnaire (CSWAL-QOL). The hypothesis of this study is that the effortful swallowing exercise would have better treatment efficacy.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with NPC
* completed radiation therapy at least 1 year
* mild to moderate swallowing disorder defined by videofluorography
* able to comply with protocal mandate, willing to perform the exercise programs, and ability to attend the weekly sessions

Exclusion Criteria:

* feeding tube insitu
* received pharyngeal surgery
* tracheostomy tube insitu
* patients who could not put effort to push posterior tongue base backward and who could not elevate their pharyngeal during swallowing
* severe swallowing disorder or aspirate defined by videofluorography
* other malignances, neurovascular disease, demyelinating disease
* cancer relapse or metastases

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in videofluoroscopic swallowing study (VFSS) | Change from Baseline in VFSS at 8 weeks
  Videofluoroscopic swallowing study (VFSS) measures the bolus transit time including: 1.oral transit time; 2. pharyngeal transit time; and 3. pharyngeal delay time. It also reveals the occurrence of swallowing aspiration or not.

SECONDARY OUTCOMES:
Change from Baseline in Chinese version of the Swallow Quality-of-Life Questionnaire (CSWAL-QOL) | Change from Baseline in CSWAL-QOL at 8 weeks
  The Chinese version of SWAL-QOL questionnaire (CSWAL-QOL) contains 10 scales related to swallowing and quality of life, including burden, eating desire, food duration, food selection, communication, fear, mental health, social functioning, sleep, and fatigue. All scales are linearly transformed into a 0-to-100 metric, with 0 indicating most dysfunction and 100 indicating no dysfunction.

OTHER OUTCOMES:
Change from Baseline in the Mann Assessment of Swallowing Ability (MASA) | Change from Baseline in MASA at 8 weeks
  The the Mann Assessment of Swallowing Ability (MASA) is designed to yield specific information about a patients's swallowing ability through examiner interpretation of responses. Two scores are obtained: a total score out of 200, and an ordinal risk rating for both aspiration and dysphagia (definite, probable, possible, unlikely).

CONTACTS AND LOCATIONS:
Overall Officials: Jenq-Yuh Ko, M.D., Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

REFERENCES:
- [Background] Hind JA, Nicosia MA, Roecker EB, Carnes ML, Robbins J. Comparison of effortful and noneffortful swallows in healthy middle-aged and older adults. Arch Phys Med Rehabil. 2001 Dec;82(12):1661-5. doi: 10.1053/apmr.2001.28006. PMID 11733879
- [Background] Huang HY, Wilkie DJ, Schubert MM, Ting LL. Symptom profile of nasopharyngeal cancer patients during radiation therapy. Cancer Pract. 2000 Nov-Dec;8(6):274-81. doi: 10.1046/j.1523-5394.2000.86007.x. PMID 11898144
- [Background] Hughes PJ, Scott PM, Kew J, Cheung DM, Leung SF, Ahuja AT, van Hasselt CA. Dysphagia in treated nasopharyngeal cancer. Head Neck. 2000 Jul;22(4):393-7. doi: 10.1002/1097-0347(200007)22:43.0.co;2-2. PMID 10862024
- [Background] Kotz T, Federman AD, Kao J, Milman L, Packer S, Lopez-Prieto C, Forsythe K, Genden EM. Prophylactic swallowing exercises in patients with head and neck cancer undergoing chemoradiation: a randomized trial. Arch Otolaryngol Head Neck Surg. 2012 Apr;138(4):376-82. doi: 10.1001/archoto.2012.187. PMID 22508621
- [Background] Ku PK, Yuen EH, Cheung DM, Chan BY, Ahuja A, Leung SF, Tong MC, van Hasselt A. Early swallowing problems in a cohort of patients with nasopharyngeal carcinoma: Symptomatology and videofluoroscopic findings. Laryngoscope. 2007 Jan;117(1):142-6. doi: 10.1097/01.mlg.0000248738.55387.44. PMID 17202944
- [Background] Kulbersh BD, Rosenthal EL, McGrew BM, Duncan RD, McColloch NL, Carroll WR, Magnuson JS. Pretreatment, preoperative swallowing exercises may improve dysphagia quality of life. Laryngoscope. 2006 Jun;116(6):883-6. doi: 10.1097/01.mlg.0000217278.96901.fc. PMID 16735913
- [Background] Lam PM, Lai CK. The validation of the Chinese version of the Swallow Quality-of-Life Questionnaire (SWAL-QOL) using exploratory and confirmatory factor analysis. Dysphagia. 2011 Jun;26(2):117-24. doi: 10.1007/s00455-010-9272-6. Epub 2010 Mar 4. PMID 20204414
- [Background] Lazarus C, Logemann JA, Song CW, Rademaker AW, Kahrilas PJ. Effects of voluntary maneuvers on tongue base function for swallowing. Folia Phoniatr Logop. 2002 Jul-Aug;54(4):171-6. doi: 10.1159/000063192. PMID 12169803
- [Background] Logemann JA. Role of the modified barium swallow in management of patients with dysphagia. Otolaryngol Head Neck Surg. 1997 Mar;116(3):335-8. doi: 10.1016/S0194-59989770269-9. PMID 9121786
- [Background] Shaker R, Easterling C, Kern M, Nitschke T, Massey B, Daniels S, Grande B, Kazandjian M, Dikeman K. Rehabilitation of swallowing by exercise in tube-fed patients with pharyngeal dysphagia secondary to abnormal UES opening. Gastroenterology. 2002 May;122(5):1314-21. doi: 10.1053/gast.2002.32999. PMID 11984518
- [Background] Tang Y, Shen Q, Wang Y, Lu K, Wang Y, Peng Y. A randomized prospective study of rehabilitation therapy in the treatment of radiation-induced dysphagia and trismus. Strahlenther Onkol. 2011 Jan;187(1):39-44. doi: 10.1007/s00066-010-2151-0. Epub 2010 Dec 10. PMID 21136031
- [Background] van der Molen L, van Rossum MA, Burkhead LM, Smeele LE, Rasch CR, Hilgers FJ. A randomized preventive rehabilitation trial in advanced head and neck cancer patients treated with chemoradiotherapy: feasibility, compliance, and short-term effects. Dysphagia. 2011 Jun;26(2):155-70. doi: 10.1007/s00455-010-9288-y. Epub 2010 Jul 11. PMID 20623305
- [Background] Wang TG, Chang YC, Chen WS, Lin PH, Hsiao TY. Reduction in hyoid bone forward movement in irradiated nasopharyngeal carcinoma patients with dysphagia. Arch Phys Med Rehabil. 2010 Jun;91(6):926-31. doi: 10.1016/j.apmr.2010.02.011. PMID 20510985
- [Background] Wu CH, Hsiao TY, Ko JY, Hsu MM. Dysphagia after radiotherapy: endoscopic examination of swallowing in patients with nasopharyngeal carcinoma. Ann Otol Rhinol Laryngol. 2000 Mar;109(3):320-5. doi: 10.1177/000348940010900315. PMID 10737318
- See also: American Speech-Language-Hearing Association — http://www.asha.org/